CLINICAL TRIAL: NCT04236154
Title: "Prescribing" Exercise to Cancer Patients At High-Risk for Falls
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Andersen Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-007775; NCI-2020-00367 (Other: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2020-01-16; First posted 2020-01-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cancer
Keywords: Exercise, Falls
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: The investigator will incrementally increase the exercise prescription for groups of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Pedometer — Participants will wear a pedometer for 4 days at baseline, and 4-6 weeks later. Baseline readings will be used to derive an individualized exercise program for each participant based on the assigned experimental arm.
Other: Actigraph — Participants will wear a Actigraph for 4 days at baseline and 4-6 weeks later. Baseline readings will be used to derive an individualized exercise program for each participant based on the assigned experimental arm.
Other: Perturbation Treadmill — Participants will walk on an instrumented treadmill while wearing a safety harness at baseline and 4-6 weeks later. The perturbation treadmill will assess an individual's risk for falling. Baseline readings will be used to derive an individualized exercise program for each participant based on the assigned experimental arm.

SUMMARY:
Falls are common and catastrophic in cancer patients. Cancer patients are vulnerable to falls due to muscle loss. In prescribing exercise in a data driven manner to cancer patients, our hypothesis is this "prescription" for exercise will eventually be demonstrated to reduce the occurrence of injurious falls.

ELIGIBILITY:
Inclusion Criteria:

* Any cancer diagnosis, as documented in medical record, other than non-melanoma skin cancer.
* No issues such as unstable angina or loss of a limb that would preclude exercise.

Exclusion Criteria:

* Diagnosis of non-melanoma skin cancer
* Unstable angina
* Loss of limb, which limits exercise capabilities at the discretion of the Principal Investigators
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
ABC Activities Specific Balance Confidence Scale (exploratory outcome) | Change from baseline ABC scale at 4-6 weeks
  Patient Reported Outcome 0% No confidence, 100% Complete Confidence, higher score= better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials